CLINICAL TRIAL: NCT00343239
Title: Docetaxel, Cisplatin and Fluorouracil Combination in the Neoadjuvant Treatment of Locally Advanced Gastric Adenocarcinoma : Phase II Clinical Study
Brief Title: Docetaxel in Locally Advanced Gastric Adenocarcinoma
Acronym: NEOTAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_00072
Record Dates: First submitted 2006-06-21; First posted 2006-06-22 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil

ARMS (1):
- Docetaxel/Cisplatin/Fluorouracil (DCF) (Experimental): DCF combination for three 21-day cycles unless a disease progression is observed at the tumor assessment scheduled after the second cycle or due to patient intolerability
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Docetaxel — Formulation: infusion solution
  Route of administration: IV infusion on the first day of each 21-day cycle
  Dose regimen: 75 mg/m2
Drug: Cisplatin — Formulation: infusion solution
  Route of administration: IV infusion on the first day of each 21-day cycle
  Dose regimen: 75 mg/m2
Drug: Fluorouracil — Formulation: infusion solution
  Route of administration: IV infusion on the first day of each 21-day cycle
  Dose regimen: 750 mg/m2/day for 5 days

SUMMARY:
Study objectives:

To determine Ro resection rate of Docetaxel, cisplatin and fluorouracil combination for the treatment of neoadjuvant gastric carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric adenocarcinoma diagnosis
* Selected Stage IIB (T3N0M0), Stage IIIA (T2aN2M0, T2bN2M0, T3N1M0, T4N0M0), Stage IIIB (T3N2M0) and selected Stage IV (all T4 , NM0, all TN3M0's). Clinical staging performed with endoscopic ultrasound and CT. Laparotomy or laparoscopy is preferred to determine resectability and peritoneal involvement.
* ECOG performance status between 0 and 2
* Acceptable hematological profile :

  * WBC (White Blood Cell) count ≥4000/mm3
  * Platelet count ≥100 000 mm3
  * Hemoglobin ≥9 g/100 mL (if lower, may be included following transfusion)
* Adequate renal function

  * Serum creatinine <1.2 mg/dl or calculated creatinine clearance in 24-hours urine >60 mL/min.
* Adequate hepatic function

  * Bilirubin < UNL
  * Transaminases (ALT, AST) <2.5 x UNL
  * Alcaline phosphatase <2.5 x UNL
* Adequate pulmonary function
* Adequate cardiac function
* No prior chemotherapy for gastric cancer

Exclusion Criteria:

* Other histological types of gastric cancer (leiomyosarcoma, lymphoma) than adenocarcinoma
* Pregnant or lactating patients
* Patients with brain, bone or other metastases; peritoneal involvement
* Other serious underlying medical conditions which could impair the ability of the patient to participate in the study (congestive heart failure, serious arrhythmia, uncontrolled diabetes mellitus, serious neuropathy), history of myocardial infarction within 6 months prior to study entry
* Previous or other current malignancies, with the exception of carcinoma of the cervix uteri or breast cancer or basal cell skin cancer and a disease-free period shorter than 5 years
* Active infection and other serious disease
* Any other experimental drugs within a 4-week period prior to the study
* Contraindications for the use of any study drug (e.g. history of hypersensitivity to the contents of the study drugs)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine the R0 resection rate for the treatment of locally advanced gastric carcinoma with Docetaxel, Cisplatin, Fluorouracil combination. | 3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Ozdemir N, Abali H, Vural M, Yalcin S, Oksuzoglu B, Civelek B, Oguz D, Bostanci B, Yalcin B, Zengin N. Docetaxel, cisplatin, and fluorouracil combination in neoadjuvant setting in the treatment of locally advanced gastric adenocarcinoma: Phase II NEOTAX study. Cancer Chemother Pharmacol. 2014 Dec;74(6):1139-47. doi: 10.1007/s00280-014-2586-6. Epub 2014 Sep 19. PMID 25234436